CLINICAL TRIAL: NCT02543996
Title: Human Biospecimen Procurement and Analysis to Support Translational Research to Identify Genetic Etiology and Disease Mechanism(s) in Rare Genetic Vascular/Cardiovascular Diseases
Brief Title: Human Biospecimen Procurement Protocol: Biorepository to Support Translational Research to Identify Disease Mechanism(s)
Status: Recruiting | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 150190; 15-H-0190
Record Dates: First submitted 2015-09-05; First posted 2015-09-09 (Estimated); Last update posted 2026-01-09 (Actual); Status verified 2026-01-07

CONDITIONS: Undiagnosed Diseases; Cardiovascular Disease
Keywords: Sample Collection; Laboratory Research Specimens; Biospecimen Procurement; Rare Diseases; Natural History
MeSH Terms: conditions — Undiagnosed Diseases; Cardiovascular Diseases; Rare Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Affected or unaffected cohorts (including genetic carriers or non-carriers as: Affected or unaffected cohorts (including genetic carriers or non-carriers as reference biospecimens)

SUMMARY:
Background:

Studies show that rare genetic variants might lead to diseases. Researchers want to collect blood and tissue samples so they can study them and better understand diseases.

Objective:

To collect blood and tissue samples for studies to identify underlying causes of disease.

Eligibility:

People of all ages

Design:

Participants will have blood and/or tissue samples collected.

Samples can be collected at the NIH Clinical Center. Participants doctors can collect the samples and send them to NIH. NIH staff can collect samples off site.

For blood samples, blood is taken from an arm vein using a needle.

Tissue collection may involve:

Buccal smear: Cells are collected by scraping the inside of the cheek with a cotton swab.

Saliva collection: Participants spit into a cup.

Skin biopsy: A special needle takes a very small skin sample.

Surgical waste tissue: If participants have surgery, NIH may receive samples of tissue that

would routinely be removed.

Umbilical cord or cord blood collection: If a participant has a baby, NIH may receive a

small piece of the umbilical cord or blood from the cord once the baby is delivered.

DETAILED DESCRIPTION:
The diversity of human research programs at the National Institutes of Health (NIH) provides a unique opportunity to study different patient populations with monogenetic and undiagnosed diseases with vascular implications. Patient populations with mutations in almost every major signaling pathway related to cardiovascular diseases are actively investigated at the NIH Clinical Center. The purpose of this protocol is to obtain and analyze human biospecimens from affected and unaffected cohorts (as reference biospecimens) to identify genetic etiology and/or underlying disease mechanism(s) in rare genetic vascular/cardiovascular conditions. The collections will consist of biospecimens obtained from participants consented under this protocol and will also provide for the continued storage and analysis of biospecimens previously obtained from NIH Institutional Review Board (IRB)-approved protocols, or from NIH protocols nearing completion. The biospecimens collected under this protocol will include blood (plasma, serum, peripheral blood mononuclear cells (PBMCs)), saliva, buccal mucosa, urine, and skin biopsies. Additional biospecimens collected under other protocols may also be transferred to this protocol, including, tissue and fluid aspirates (cerebrospinal fluid, ascites, etc.), bone marrow, urine, saliva, skin biopsies, surgical tissue waste, malignant and non-malignant tissue samples, and/or other direct derivatives from human tissues (i.e. DNA, RNA, and induced pluripotent stems cells). Post-delivery umbilical cord core blood and cord tissue waste will be collected at the time of delivery under this protocol and/or shared if obtained under other protocols. Biospecimens may also be obtained as shared samples of clinically indicated procedures done inside or outside NIH, provided the subject consents to this protocol.

The primary objective of this protocol is to create a robust resource to support basic and translational research by providing a mechanism for collecting, tracking, storing, dispensing, analyzing, and disposing of laboratory research samples from affected and unaffected cohorts. This research will advance high-quality research in the areas of genetics and personalized medicine.

As this is not a treatment protocol, there is no primary endpoint. Research studies will include, but not be limited to, genomic studies, primary cell isolation and cell culture studies for molecular and biochemical analysis, immunohistological analysis, generation of patient-specific in vitro disease models (i.e. IPSCs), etc. As science is a continuously evolving field, technological advances in research methods will be incorporated into research studies accordingly.

ELIGIBILITY:
* INCLUSION CRITERIA (SUBJECTS MUST MEET ONE OF THE FOLLOWING):
* Age: older than 1 month of age
* Affected pregnant women if they have been referred with a known or suspected pathology or if they become pregnant while on study.
* Unaffected related pregnant women (including spouses/partners) for cord blood and tissue collection (surgical waste) only at the time of delivery.
* Cognitively impaired individuals that are affected
* Cognitively impaired individuals that are related to an affected subject.
* Subjects willing to provide informed consent.

EXCLUSION CRITERIA:

* Healthy volunteers unable to give informed consent
* Cognitively impaired individuals who are not affected
* Cognitively impaired individuals who are not related to affected subjects.

Ages: 1 Month to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Affected or unaffected cohorts (including genetic carriers or non-carriers as reference biospecimens)
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2015-09-17 (Actual); Primary Completion 2040-06-04 (Estimated); Study Completion 2050-05-22 (Estimated)

PRIMARY OUTCOMES:
To procure human biospecimens from affected and unaffected cohorts for on-going and future basic and translational research studies to identify underlying disease mechanism(s) | ongoing
  The primary objective is to procure human biospecimens from affected and unaffected cohorts for on-going and future basic translational research studies to identify underlying disease mechanism(s) and potential therapeutic approaches

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Boehm, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2015-H-0190.html